CLINICAL TRIAL: NCT01916746
Title: Safety and Effectiveness of Transvaginal Resection of Pregnancy Tissue in the Treatment of Caesarean Scar Pregnancy
Brief Title: Treatment of Caesarean Scar Pregnancy
Acronym: CSP
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Shu-Qin Chen (Other)
Responsible Party: Sponsor-Investigator, Shu-Qin Chen, associate professor of gynaecology and obstetrics, First Affiliated Hospital, Sun Yat-Sen University
Organization: First Affiliated Hospital, Sun Yat-Sen University (Other)
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: CHEN-CSP; CSP-2013 (Other: Hospital Ethical Committee)
Record Dates: First submitted 2013-07-25; First posted 2013-08-06 (Estimated); Last update posted 2013-08-06 (Estimated); Status verified 2013-01

CONDITIONS: Caesarean Scar Pregnancy
Keywords: Caesarean Scar Pregnancy; Transvaginal Resection; treatment

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- transvaginal resection of pregnancy tissue (Experimental)
  Interventions: Procedure: transvaginal resection of pregnancy tissue

INTERVENTIONS:
Procedure: transvaginal resection of pregnancy tissue — Patient were under general anaesthesia, placed in a dorsal lithotomy position and the bladder emptied. Expose, grasp and traction the cervix. And adrenaline (600 ug/l; 10-20 ml) was injected submucosally at the level of the cervicovaginal junction. An incision was made at the anterior cervicovaginal junction, and the bladder was dissected away until the anterior peritoneal reflection was identified. The anterior drawing hook was inserted into the vaginal incision to retract the bladder upwards. The CSP was identified as a'purple bulge' located in the anterior part of the lower uterine segment. A transverse incision was made over the most prominent area of the bulge. Ectopic pregnancy tissue inside the bulge was removed, and suction curettage through the incision on the uterus isthmus was subsequently performed. The edges of the incision were trimmed with scissors, and the myometrial and vaginal defects were closed with a continuous locking suture using 2-0 absorbable sutures.

SUMMARY:
The aim of this study is to further demonstrate the safety and effectiveness of transvaginal resection of pregnancy tissue in the treatment of Caesarean Scar Pregnancy (CSP).

ELIGIBILITY:
Inclusion Criteria:

* pre-operative diagnosed as CSP
* hemodynamic stability

Exclusion Criteria:

* cervical pregnancy
* incomplete abortion
* gestational trophoblastic disease
* diagnosis unidentified

Sex: Female | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 150 (Estimated)
Dates: Start 2013-01; Primary Completion 2015-12 (Estimated)

PRIMARY OUTCOMES:
The safety of transvaginal resection of pregnancy tissue in the treatment of CSP. | one week
  index of blood loss, haemoglobin decrease(post-operation day 2 minus pre-operation), operation time, perioperation complications,change to other treatment procedure are collected to evaluate the safety of this procedure.
the effectiveness of transvaginal resection of pregnancy tissue in the treatment of CSP. | six months
  serum hCG are measured every week till post-operation till it resolute to normal level. and transvaginal ultrasound are performed every month post-operation till there is no sign of any pregnancy residues.

SECONDARY OUTCOMES:
Baseline clinical characteristic of patient when diagnosed with CSP | one week
  age, gravity and parity, previous caesarean section times, interval from last caesarean section, gestation age when diagnosed, pre-treatment human chorionic gonadotropin(hCG) level and ultrasound characteristic details are collected to investigate the relation between these index and CSP
three year recurrence rate | three years after the procedure
  the following pregnancy result of patient are inquired every year till three years post-operative to evaluate the influence of this procedure on further pregnancy.

CONTACTS AND LOCATIONS:
Overall Officials: Chen Shu-Qin, M.D&PhD., Study Director — First Affiliated Hospital, Sun Yat-Sen University; Li Jin-Bo, M.D, Principal Investigator — First Affiliated Hospital, Sun Yat-Sen University; Yao Shu-Zhong, M.D&Ph.D, Study Chair — First Affiliated Hospital, Sun Yat-Sen University
Locations (1):
- The First Affiliated Hospital of Sun Yat-sen University, Guangzhou, Guangdong, China